CLINICAL TRIAL: NCT01416324
Title: A First Time in Human, Single Blind, Randomized, Placebo-controlled,Dose Escalating Crossover Study to Evaluate the Safety,Tolerability, Pharmacokinetic and Pharmacodynamic Parameters of Single Doses of GSK2330672 in Healthy Volunteers
Brief Title: First Time in Human Study Using GSK2330672
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 114985
Record Dates: First submitted 2011-06-16; First posted 2011-08-15 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: pharmacodynamics; first time in human; pharmacokinetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-((((3R,5R)-3-butyl-3-ethyl-7-(methyloxy)-1,1-dioxido-5-phenyl-2,3,4,5-tetrahydro-1,4-benzothiazepin-8-yl)methyl)amino)pentanedioic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK2330672 (Experimental): experimental study drug
  Interventions: Drug: 0.1 mg GSK2330672; Drug: 0.3 mg GSK2330672; Drug: 1 mg GSK2330672; Drug: 3 mg GSK2330672; Drug: 10 mg GSK2330672; Drug: 30 mg GSK2330672; Drug: 60 mg GSK2330672
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — Vehicle used to dilute the powder for oral administration.
  Arms: Placebo
Drug: 0.1 mg GSK2330672 — GSK2330672 is available as a white to almost white solid powder diluted in vehicle for oral administration.
  Arms: GSK2330672
Drug: 0.3 mg GSK2330672 — GSK2330672 is available as a white to almost white solid powder diluted in vehicle for oral administration.
  Arms: GSK2330672
Drug: 1 mg GSK2330672 — GSK2330672 is available as a white to almost white solid powder diluted in vehicle for oral administration.
  Arms: GSK2330672
Drug: 3 mg GSK2330672 — GSK2330672 is available as a white to almost white solid powder diluted in vehicle for oral administration.
  Arms: GSK2330672
Drug: 10 mg GSK2330672 — GSK2330672 is available as a white to almost white solid powder diluted in vehicle for oral administration.
  Arms: GSK2330672
Drug: 30 mg GSK2330672 — GSK2330672 is available as a white to almost white solid powder diluted in vehicle for oral administration.
  Arms: GSK2330672
Drug: 60 mg GSK2330672 — GSK2330672 is available as a white to almost white solid powder diluted in vehicle for oral administration.
  Arms: GSK2330672

SUMMARY:
The purpose of this study is to look at the safety and tolerability of increasing single doses of GSK2330672 in healthy volunteers.

DETAILED DESCRIPTION:
This is a single blind, randomized, placebo-controlled, dose escalating, crossover, first time in human study to examine safety, tolerability, pharmacokinetic and pharmacodynamic parameters of GSK233672. Single blind indicates that the subjects and investigator are blinded to treatment but the GSK study team could be unblinded for ongoing review of interim safety data required for dose escalation.

Subjects will participate in 4 dosing periods. Subjects will enter the clinic prior to dinner time on the evening of Day -1 of each period and will remain in residence through the morning of Day 3. Barring any safety or tolerability concerns, subjects will be released at this time provided they have had at least 1 bowel movement after dosing in the clinic.

Subjects will return for their next scheduled dosing period. This process will be repeated for each dosing period. Subjects will return approximately 1 week after check out from their last dosing period for a follow up visit. Subjects will receive standardized meals meeting specific criteria starting with dinner on Day-1 and continuing through Day 1. Standard meals will be provided for the remainder of their stay in the clinic. After an overnight fast, subjects will take their study drug on the morning of Day 1. Dosing will be followed by breakfast and frequent blood sampling to assess pharmacokinetic and pharmacodynamic parameters. Scheduled assessments of heart rate, blood pressure, respiratory rate, ECGs, and clinical laboratories will be obtained to monitor subject safety. Subjects will be connected to cardiac telemetry monitors and will periodically undergo spirometry testing of ventilation parameters. Stool form and frequency of bowel movements will be recorded. All fecal samples will be collected from participants for 48 hours after dosing of study drug, or until they have had at least 1 bowel movement after dosing, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer
* 18-60 yrs of age
* for subjects age 50 and above: negative fecal occult blood test within 3 months prior to expected start of dosing, and normal results from sigmoidoscopy or colonoscopy within 5 yrs prior to dosing.
* if female, must be of non-childbearing potential

Exclusion Criteria:

* pregnant or breastfeeding females
* positive HIV
* positive Hep B, or Hep C within 3 months of screening
* positive drugs of abuse screening
* triglycerides > 250 mg/dL
* current or chronic history of liver disease
* any gastrointestinal or gastrointestinal related conditions that could affect fat or bile acid reabsorption
* pancreatitis
* colon cancer or 1st degree relative who has had colon cancer
* abnormal lung function tests
* inability to perform lung function tests
* unwilling to abstain from smoking, alcohol, caffeine, illicit drugs as directed by the site staff
* exposure to more than 4 new chemical entities in the 12 months prior to the first dosing day.
* where participation in the study would results in donation of more than approximately 550mL of blood in a 56-day period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2011-06-15 (Actual); Primary Completion 2011-09-09 (Actual); Study Completion 2011-09-09 (Actual)

PRIMARY OUTCOMES:
Change in vital signs | 1, 2, 4, 8, 12, 24, 48 hours
  frequency and absolute value change in heart rate, blood pressure, respiration rate relative to placebo
ECGs relative to placebo | 1, 2, 4, 8, 12, 24, 48 hours
  frequency of clinically significant changes in 12-lead ECG parameters relative to placebo
Changes in clinical lab results | 24 hours
  Changes in clinical chemistry, hematology, urinalysis results relative to placebo
lung function tests | 1, 3, 8, 24 hours
  Measure changes in FEV, FVC, FEF 25-75%, PEFR relative to placebo
Adverse events relative to placebo | 48 hour monitoring
  Frequency and severity of adverse events relative to placebo

SECONDARY OUTCOMES:
Measurement of the maximum concentration (Cmax) for study drug | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3.5, 5, 6.5, 8, 9.5, 12.5 hours
Measurement of the time to achieve maximum concentration (tmax) for study drug | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3.5, 5, 6.5, 8, 9.5, 12.5 hours
Measurement of area under the curve (AUC) for study drug | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3.5, 5, 6.5, 8, 9.5, 12.5 hours
Measurement of half life (t 1/2) of study drug | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3.5, 5, 6.5, 8, 9.5, 12.5 hours
Measurement of apparent clearance (CL/F) of the study drug | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3.5, 5, 6.5, 8, 9.5, 12.5 hours
Measurement of the apparent volume of distribution (V/F) of the study drug | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3.5, 5, 6.5, 8, 9.5, 12.5 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 114985 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/114985?search=study&search_terms=114985#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 114985 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114985 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114985 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114985 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114985 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114985 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114985 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register